A Multimethod Evaluation of Tobacco Treatment Trial Recruitment Messages for Current Smokers Recently Diagnosed With Cancer: Pilot Factorial Randomized Controlled Trial

NCT #: N/A

Document Date: 11/19/2020

## **Information Sheet**

Please read this consent document carefully before you decide to participate in this study.

**Purpose of the Study:** Welcome to the United States Healthy Living Survey. We are conducting this study to find out how people aged 18 and over make decisions about their health. By the end of this study, we hope to identify what types of information are most helpful for people to make better decisions about their health behaviors, such as smoking.

Time required: 15-20 minutes.

**Risks and Benefits:** There are no direct benefits to you for participating in the study. There will be no potential risk for physical, psychological or economic harm.

**Compensation**: You will receive compensation for your participation. The panel company you are working with will arrange payment once you have finished the survey. Successful completion of this survey will result in a nominal reimbursement of less than \$5.

**Confidentiality:** There is a minimal risk that security of any online data may be breached, but since no identifying information will be collected, and the online host (Qualtrics) uses several forms of encryption, it is unlikely that a security breach of the online data will result in any adverse consequence for you.

**Voluntary participation:** Your participation in this study is completely voluntary. There is no penalty for not participating, and you do not have to answer any question you do not wish to answer.

**Right to withdraw from the study:** You have the right to withdraw from the study at any time without consequence.

Whom to contact if you have questions about the study:

## Elyse R. Park, Ph.D., MPH

Associate Professor of Psychiatry, Harvard Medical School | Mongan Institute for Health Policy Center Massachusetts General Hospital | 50 Staniford Street | Room 907 | Boston, MA 02114 Research Tel: 617.724.6836 | Research Fax: 617.;724.4738 | Clinical Tel: 617.643.7257 Email: epark@mgh.harvard.edu

## Jordan M. Neil, Ph.D.

Postdoctoral Research Fellow
Harvard Medical School | Mongan Institute Health Policy Center
Massachusetts General Hospital | 100 Cambridge Street | Suite 1600 | Boston, MA 02114
Research Tel: 617-643-5165
Email: jmneil@mgh.harvard.edu

## Whom to contact about your rights as a research participant in the study:

Partners Human Research Committee, 399 Revolution Drive, Suite # 710, Somerville MA, 02145; phone 857-282-1900.

- □ Yes Please proceed to the survey.
- □ No Thank you for your time.